CLINICAL TRIAL: NCT03282552
Title: High Flow Oxygen Therapy Versus Conventional Oxygen Therapy in Cardiac Surgery Patients-OPTICAR Study
Brief Title: High Flow Oxygen Therapy Versus Conventional Oxygen Therapy in Cardiac Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Stavros Theologou, Principal Investigator, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NKU Athens
Record Dates: First submitted 2017-08-01; First posted 2017-09-14 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Group 1 (Active Comparator): The intervention consists of the implementation of Nasal Cannula High Flow Oxygenation as an oxygen treatment at Study Group 1, whereas oxygen supply was provided via Venturi mask at the standard oxygen patients' treatment.
  The first Study Group will include patients on Nasal Cannula High Flow Oxygenation with initial settings of FiO2=60% and gas flow=60L/min.
  Interventions: Device: Nasal Cannula High Flow Oxygen
- Study Group 2 (Active Comparator): The intervention consists of the implementation of Nasal Cannula High Flow Oxygenation as an oxygen treatment at Study Group 2, whereas oxygen supply was provided via Venturi mask at the standard oxygen patients' treatment.
  The second Study Group will include patients on Nasal Cannula High Flow Oxygenation with initial settings of FiO2=60% and gas flow=40L/min.
  Interventions: Device: Nasal Cannula High Flow Oxygen
- Control group (No Intervention): In the third group (control group) all patients will receive oxygen treatment according to the standard practice of our cardiac ICU department, i.e., Venturi mask with FiO2=60% and flow of 15L/min.
  In this group all patients will receive the usual standard of care, with no other interventions included

INTERVENTIONS:
Device: Nasal Cannula High Flow Oxygen — Nasal Cannula High Flow Oxygenation will be implemented at these study groups . (1st study group, and 2nd study group)
  Arms: Study Group 1; Study Group 2

SUMMARY:
High flow oxygen therapy has been applied after extubation in cardiac surgery patients with uncertain efficacy. The current authors plan to conduct a prospective, randomized, controlled study of nasal high flow therapy (NHF) application with high (60L/min) or low flow (40L/min) oxygen mixture administration versus standard oxygen treatment (Venturi mask) after extubation of patients undergoing elective or non-elective cardiac surgery.

DETAILED DESCRIPTION:
Over the past decade, nasal high flow (NHF) has been introduced for oxygen therapy in adults. Its indications have been expanded, especially in cases of acute hypoxemic respiratory failure.

The device consists of an air/oxygen blender connected via an active heated humidifier to a nasal cannula, through a single limb, heated inspiratory circuit. It delivers a fraction of inspired oxygen (FiO2) from 21% to 100% with a flow rate up to 60 L/min. FiO2 adjustments are independent of the set flow rate so that the patient is given heated, humidified high-flow oxygen, with a flow that can be adjusted above the patient's maximum inspiratory flow rate, thereby increasing confidence about the actual FiO2 being delivered to the patient. These device characteristics make it more promising in comparison with conventional low- and high-flow oxygen devices (e.g., nasal cannula, non-rebreathing masks, Venturi masks), especially in patients with high inspiratory flow rates, such as patients with acute respiratory failure (ARF).

The benefits arising from application of oxygen with high flow rates via NHF are

1. reduction in the entrainment of room air and thus ensuring higher and more stable FiO2 values,
2. generation of positive airway pressures during expiration as a result of the expiratory resistance imposed to the patient's exhalation against the continuous high flow of incoming oxygen gas,
3. improving mucociliary function and clearance of secretion by continuous heating and humidifying of the administered gas,
4. reducing dead space ventilation and
5. reducing work of breathing. All the aforementioned NHF mechanisms of actions exert various effects on the respiratory system, including improved gas exchange, lower respiratory rate and effort and improved lung mechanics which are correlated with more comfort and less subjective dyspnea.

Respiratory complications after cardiac surgery can affect morbidity and mortality, and increase the healthcare cost. Advanced age, duration of extracorporeal circulation, history of significant underlying cardiac or pulmonary disease and phrenic nerve injury are the main prognostic factors for post cardiac surgery respiratory complications.

Traditionally, low- and high-flow oxygen systems are used to reverse postsurgical respiratory complications with or without addition of continuous (CPAP) or bi-level (NIV) positive airway pressure.

NHF might be superior for the prevention or treatment of those respiratory complications, since it can provide high-flow of heated and hydrated oxygen while the positive airway pressure created by the high gas flow can recruit alveoli and increase the end-expiratory lung volume.

Studies applying NHF immediately after extubation in cardiac surgery patients revealed better oxygenation and less need for advanced methods of respiratory support compared to conventional oxygen devices , and similar results compared to noninvasive ventilation. However, Zochios et al, summarized all the available up to date data of NHF compared to conventional oxygen devices and non-invasive ventilation in patients undergoing cardiothoracic surgery and they did not find any further benefit by NHF use. The aforementioned discrepancy could be explained by the differences in the studied populations and NHF flow settings. The proposed initial flow rate differs among the studies, with some authors suggesting initial lower flows (35-40 L/min) that will be better tolerated by the patients and others suggesting initial maximal flows (60 L/min) to rapidly relieve dyspnea and prevent muscle fatigue.

Aim The primary goal of the study is to evaluate the efficacy of NHF (with initial flows of 60 L/min or 40 L/min) versus conventional oxygen systems on respiratory parameters (respiratory rate, pO2/ FiO2, spO2, use of accessory muscles, dyspnoea, comfort and tolerance by using the visual analogue scale) immediately after the extubation of cardiac surgery patients.

Additional goals of the study are to compare two different initial NHF flows of 60 L/min and 40 L/min, ICU Length of Stay, Hospital Length of Stay, rates of ICU re-admission and re-intubation and any other respiratory / non-respiratory complications and adverse events. Moreover, the rate of failure of the initial treatment will be recorded (as a major measure of treatment efficacy).

Method

This is a prospective, non-blinded, randomized study in post-extubated cardiac surgery patients. The study population will consist of three patient groups:

The first group (Study Group 1) will include patients on NHF with initial settings of FiO2=60% and gas flow=60L/min.

The second group (Study Group 2) will include patients on NHF with initial settings of FiO2=60% and gas flow=40L/min In the third group (control group) all patients will receive oxygen therapy according to the standard practice of our cardiac ICU department, i.e., Venturi mask with FiO2=60% and flow of 15L/min.

Patients in both study groups would be weaned off the NHF as follows; First reducing FiO2 gradually to 50%, and then gradually reducing the gas flow (either from 60l/min or 40/min, depending on the study group) down to 30l/min, aiming at the final wean-off goal of 20l/min, unless the attending physician decides to wean-off patient to Venturi mask directly from a higher gas flow supply (e.g.: 30-25l/min) Treatment failure will be defined as any crossover from one treatment to another due to patient's respiratory distress and discomfort. To be more specific, switch of gas flow from 40L/min to 60L/min, crossover from either NHF group to standard practice (Venturi mask) or need for more advanced respiratory support such as non-invasive ventilation or invasive mechanical ventilation.

Any implemented treatment would also be defined as "failure" when any irreversible (for at least 48 hours) FiO2/gas-mixture flow escalation might be needed, either it is being recorded on Study group 1 & 2 or Control group.

An initial power analysis was based on a predicted, average failure rate of 15% in the 2 NHF groups and a failure rate of 51% in the control group; this analysis yielded the need for enrollment of a total of 41 NHF patients and 21 controls for alpha = 0.05 and power=0.80. To ensure equal numbers of patients in each one of the 2 NHF groups, the authors decided to actually enroll 42 NHF patients (n=21 for each NHF group) and 21 controls, resulting in a total enrollment of 63 patients. At one year after study initiation, actual, total enrollment amounted to 45 patients. At this time point, the Data Monitoring Committee (after confirming the safe application of the study protocol) recommended the continuation of the study until the enrollment of 99 patients (n=33 for each one of the 3 groups); the rationale for this was to compensate for possible dropouts and/or missing data (especially for the secondary and "other" outcomes). Accordingly, the study was completed with an actual enrollment of 99 patients.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac ICU adult patients
* >18 years
* After elective or urgent cardiac surgery
* Successful Spontaneous Breathing Trial (SBT) with T-piece and FiO2=60%.
* pO2/ FiO2 <200
* Hemodynamically stable (160>SAP>90mmHg)

Exclusion Criteria:

* Obstructive Sleep Apnea Syndrome supported by CPAP
* COPD, officially diagnosed, respiratory failure with serum blood ph <7,35.
* Patients with tracheostomy,
* DNR status,
* Glasgow Coma Scale score < 13,
* Insufficient knowledge of Greek Language
* Visual or hearing impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Successful weaning (i.e. absence of treatment failure) from Nasal Cannula High Flow Oxygenation post extubation from cardiac surgery within at least 48 hours | Up to at least 48 hours post extubation or until ICU discharge (predicted cardiothoracic ICU stay could occasionally extend up to 7 days)
  Successful weaning (i.e. absence of treatment failure as further described in methods) would be defined as = 0 when there would be avoided successfully any alternation with other mode of oxygen therapy, or re-intubation, or Non Invasive Ventilation.
  For all groups: Unsuccessful weaning (i.e. actual treatment failure as further described in methods) would be defined as =1 when there would not be avoided any alternation with other oxygen therapy, re-intubation, Non Invasive Ventilation

SECONDARY OUTCOMES:
Successful maintenance of Respiration rate within normal range (12-20/min) on initial air flow at 60 L/min with Nasal Cannula High Flow Oxygenation | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  Successful maintenance of Respiratory rate within normal range would be defined as = 0. Unsuccessful (=1) if exceeds normal range (12-20/min).
  Continuous monitoring and recording of implementation of air flow at 60L/min with Nasal Cannula High Flow Oxygenation
Successful maintenance of Respiration rate within normal range (12-20/min) on initial air flow of 40 L/min with Nasal Cannula High Flow Oxygenation | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  Successful maintenance of Respiratory rate within normal range would be defined as = 0. Unsuccessful (=1) if exceeds normal range (12-20/min).
  Continuous monitoring and recording of implementation of air flow at 40L/min with Nasal Cannula High Flow Oxygenation
Successful maintenance of Respiration rate within normal range (12-20/min) with Venturi mask , FiO2: 60%, 15L/min | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  Successful maintenance of Respiration rate within normal range (12-20/min) with Venturi mask , FiO2: 60%, 15L/min Continuous monitoring and recording of implementation of Venturi mask 60% fiO2, 15l/min
Recording of pO2/FiO2 ratio with initial air flow at 60 L/min with Nasal Cannula High Flow Oxygenation | Post extubation period up to 48 hours or ICU discharge
  Continuous monitoring of implementation initial air flow at 60 L/min with Nasal Cannula High Flow Oxygenation
Recording of pO2/FiO2 ratio with initial air flow at 40 L/min with Nasal Cannula High Flow Oxygenation | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  Continuous monitoring of implementation initial air flow at 40 L/min with Nasal Cannula High Flow Oxygenation
Recording of pO2/FiO2 ratio with Venturi mask FiO2: 60%, 15L/min | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  Continuous monitoring of implementation Venturi mask, FiO2: 60%, 15L/min
Successful maintenance of saturation O2 in Hemoglobulin within normal range with initial air flow at 60 L/min with Nasal Cannula High Flow Oxygenation | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  Successful maintenace of saturation O2 in Hemoglobulin > 92% would be defined as = 0.
  If saturation O2 < 92 %, then it would be definded as Unsuccessful = 1 Continuous monitoring and recording of implementation initial air flow at 60 L/min with Nasal Cannula High Flow Oxygenation
Successful maintenance of saturation O2 in Hemoglobulin within normal range with initial air flow at 40 L/min with Nasal Cannula High Flow Oxygenation | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  Successful maintenance of saturation O2 in Hemoglobulin within normal range would be defined as = 0.
  If saturation O2 < 92 %, then it would be definded as Unsuccessful = 1
  Continuous monitoring and recording of implementation initial air flow at 40 L/min with Nasal Cannula High Flow Oxygenation
Successful maintenance of saturation O2 in Hemoglobulin within normal range with Venturi mask, FiO2: 60%, 15L/min | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  Successful maintenance of saturation O2 in Hemoglobulin > 92% would be defined as = 0. If saturation O2 < 92 %, then would be defined as Unsuccessful = 1 .
  Continuous monitoring and recording of implementation Venturi mask FiO2 : 60%, 15L/min.
Mobilization of accessory respiratory muscles with initial air flow at 60 L/min with Nasal Cannula High Flow Oxygenation | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  Success would be defined as = 0 when there would be no mobilization of accessory respiratory muscles. Failure would be defined as = 1 when there would be recorded any mobilization and use of accessory respiratory muscles
Mobilization of accessory respiratory muscles with initial air flow at 40 L/min with Nasal Cannula High Flow Oxygenation | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  Success would be defined as = 0 when there would be no mobilization of accessory respiratory muscles. Failure would be defined as = 1 when there would be recorded any mobilzation and use of accessory respiratory muscles
Mobilization of accessory respiratory muscles with Venturi mask, FiO2: 60%, 15L/min To record any use of accessory respiratory muscles with Venturi mask , FiO2: 60%, 15L/min | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  Success would be defined as = 0 when there would be no mobilization of accessory respiratory muscles. Failure would be defined as = 1 when there would be recorded any mobilzation and use of accessory respiratory muscles
Comfort and tolerance of treatment with Visual Analogue Scale with initial air flow at 60 L/min with Nasal Cannula High Flow Oxygenation | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  To monitor and record comfort of patient with the diagnostic tool of Visual Analogue Scale
Comfort and tolerance of treatment with Visual Analogue Scale with initial air flow at 40 L/min with Nasal Cannula High Flow Oxygenation | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  To monitor and record comfort of patient with the diagnostic tool of Visual Analogue Scale
Comfort and tolerance of treatment with Visual Analogue Scale with Venturi mask , FiO2: 60%, 15L/min | Post extubation period up to 48 hours or ICU discharge (if cardiothoracic ICU stay was <48 hours)
  To monitor and record comfort of patient with the diagnostic tool of Visual Analogue Scale

OTHER OUTCOMES:
Length of Stay in the ICU | Post cardiothoracic ICU admission period up to 48 hours or untiI actual cardiothoracic ICU discharge
  There will be recorded the total length of stay in the ICU since admission post surgery
Length of Stay in the Hospital | Post ICU admission period up to actual hospital discharge
  There will be recorded the total length of stay in the hospital since ICU admission
Number of participants with death in the cardiothoracic ICU post extubation | Post cardiothoracic ICU admission period up to 48 hours or untiI actual cardiothoracic ICU discharge
  There will be recorded the number of participants that will pass away post extubation in the ICU
Number of participants with death in the hospital post ICU discharge | Post ICU discharge period up to actual hospital discharge
  There will be recorded the number of participants that will pass away post extubation in the hospital , after the ICU discharge
Number of participants with Atrial Fibrillation in the ICU post extubation | Post ICU admission period up to 48 hours or actual ICU discharge
  There will be recorded the number of participants that will present Atrial Fibrillation post extubation in the ICU
Number of participants with any Adverse Events in the ICU | Post cardiothoracic ICU admission period up to 48 hours or untiI actual cardiothoracic ICU discharge
  There will be recorded the number of participants that will present any Adverse Events (respiratory , non-respiratory) post extubation in the ICU
Number of participants with any Adverse Events in the Hospital | Up to 1 month, or until actual hospital discharge
  There will be recorded the number of participants that will present any Adverse Events (respiratory, non-respiratory) post extubation in the ICU, until hospital discharge.
Percentage of participants presenting unsuccessful (failed) implementation of NHFO treatment | Post cardiothoracic ICU admission period up to 48 hours or untiI actual cardiothoracic ICU discharge
  There will be recorded the number of participants that will present failure to comply with the treatment due to failing to maintain their respiratory parameters within normal range, or due to presenting intolerance and discomfort to the implementation of NHFO treatment
Number of participants with re-intubation in the ICU | Post cardiothoracic ICU admission period up to 48 hours or untiI actual cardiothoracic ICU discharge
  There will be recorded the number of participants that will be re-intubated due to deterioration of their respiratory parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Spiros Zakynthinos, Professor, Study Chair — National and Kapodistrian University of Athens; Spiridon Mentzelopoulos, AssProfessor, Study Director — National and Kapodistrian University of Athens
Locations (1):
- Evangelismos General Hospital of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pellegrini JA, Moraes RB, Maccari JG, de Oliveira RP, Savi A, Ribeiro RA, Burns KE, Teixeira C. Spontaneous Breathing Trials With T-Piece or Pressure Support Ventilation. Respir Care. 2016 Dec;61(12):1693-1703. doi: 10.4187/respcare.04816. Epub 2016 Sep 6. PMID 27601720
- [Result] Chanques G, Riboulet F, Molinari N, Carr J, Jung B, Prades A, Galia F, Futier E, Constantin JM, Jaber S. Comparison of three high flow oxygen therapy delivery devices: a clinical physiological cross-over study. Minerva Anestesiol. 2013 Dec;79(12):1344-55. Epub 2013 Jul 15. PMID 23857440
- [Result] Spoletini G, Alotaibi M, Blasi F, Hill NS. Heated Humidified High-Flow Nasal Oxygen in Adults: Mechanisms of Action and Clinical Implications. Chest. 2015 Jul;148(1):253-261. doi: 10.1378/chest.14-2871. PMID 25742321
- [Result] Ritchie JE, Williams AB, Gerard C, Hockey H. Evaluation of a humidified nasal high-flow oxygen system, using oxygraphy, capnography and measurement of upper airway pressures. Anaesth Intensive Care. 2011 Nov;39(6):1103-10. doi: 10.1177/0310057X1103900620. PMID 22165366
- [Result] Gotera C, Diaz Lobato S, Pinto T, Winck JC. Clinical evidence on high flow oxygen therapy and active humidification in adults. Rev Port Pneumol. 2013 Sep-Oct;19(5):217-27. doi: 10.1016/j.rppneu.2013.03.005. Epub 2013 Jul 8. PMID 23845744
- [Result] Parke R, McGuinness S, Eccleston M. Nasal high-flow therapy delivers low level positive airway pressure. Br J Anaesth. 2009 Dec;103(6):886-90. doi: 10.1093/bja/aep280. Epub 2009 Oct 20. PMID 19846404
- [Result] Groves N, Tobin A. High flow nasal oxygen generates positive airway pressure in adult volunteers. Aust Crit Care. 2007 Nov;20(4):126-31. doi: 10.1016/j.aucc.2007.08.001. Epub 2007 Oct 10. PMID 17931878
- [Result] Parke RL, Eccleston ML, McGuinness SP. The effects of flow on airway pressure during nasal high-flow oxygen therapy. Respir Care. 2011 Aug;56(8):1151-5. doi: 10.4187/respcare.01106. Epub 2011 Apr 15. PMID 21496369
- [Result] Parke RL, McGuinness SP. Pressures delivered by nasal high flow oxygen during all phases of the respiratory cycle. Respir Care. 2013 Oct;58(10):1621-4. doi: 10.4187/respcare.02358. Epub 2013 Mar 19. PMID 23513246
- [Result] Chikata Y, Izawa M, Okuda N, Itagaki T, Nakataki E, Onodera M, Imanaka H, Nishimura M. Humidification performance of two high-flow nasal cannula devices: a bench study. Respir Care. 2014 Aug;59(8):1186-90. doi: 10.4187/respcare.02932. PMID 24368861
- [Result] Hasani A, Chapman TH, McCool D, Smith RE, Dilworth JP, Agnew JE. Domiciliary humidification improves lung mucociliary clearance in patients with bronchiectasis. Chron Respir Dis. 2008;5(2):81-6. doi: 10.1177/1479972307087190. PMID 18539721
- [Result] Moller W, Celik G, Feng S, Bartenstein P, Meyer G, Oliver E, Schmid O, Tatkov S. Nasal high flow clears anatomical dead space in upper airway models. J Appl Physiol (1985). 2015 Jun 15;118(12):1525-32. doi: 10.1152/japplphysiol.00934.2014. PMID 25882385
- [Result] Moller W, Feng S, Domanski U, Franke KJ, Celik G, Bartenstein P, Becker S, Meyer G, Schmid O, Eickelberg O, Tatkov S, Nilius G. Nasal high flow reduces dead space. J Appl Physiol (1985). 2017 Jan 1;122(1):191-197. doi: 10.1152/japplphysiol.00584.2016. Epub 2016 Nov 17. PMID 27856714
- [Result] Mauri T, Turrini C, Eronia N, Grasselli G, Volta CA, Bellani G, Pesenti A. Physiologic Effects of High-Flow Nasal Cannula in Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2017 May 1;195(9):1207-1215. doi: 10.1164/rccm.201605-0916OC. PMID 27997805
- [Result] Lenglet H, Sztrymf B, Leroy C, Brun P, Dreyfuss D, Ricard JD. Humidified high flow nasal oxygen during respiratory failure in the emergency department: feasibility and efficacy. Respir Care. 2012 Nov;57(11):1873-8. doi: 10.4187/respcare.01575. Epub 2012 Mar 13. PMID 22417844
- [Result] Frizzola M, Miller TL, Rodriguez ME, Zhu Y, Rojas J, Hesek A, Stump A, Shaffer TH, Dysart K. High-flow nasal cannula: impact on oxygenation and ventilation in an acute lung injury model. Pediatr Pulmonol. 2011 Jan;46(1):67-74. doi: 10.1002/ppul.21326. Epub 2010 Nov 23. PMID 21171186
- [Result] Ferreyra G, Long Y, Ranieri VM. Respiratory complications after major surgery. Curr Opin Crit Care. 2009 Aug;15(4):342-8. doi: 10.1097/MCC.0b013e32832e0669. PMID 19542885
- [Result] Dimick JB, Chen SL, Taheri PA, Henderson WG, Khuri SF, Campbell DA Jr. Hospital costs associated with surgical complications: a report from the private-sector National Surgical Quality Improvement Program. J Am Coll Surg. 2004 Oct;199(4):531-7. doi: 10.1016/j.jamcollsurg.2004.05.276. PMID 15454134
- [Result] Ji Q, Mei Y, Wang X, Feng J, Cai J, Ding W. Risk factors for pulmonary complications following cardiac surgery with cardiopulmonary bypass. Int J Med Sci. 2013 Sep 10;10(11):1578-83. doi: 10.7150/ijms.6904. eCollection 2013. PMID 24046535
- [Result] Weissman C. Pulmonary complications after cardiac surgery. Semin Cardiothorac Vasc Anesth. 2004 Sep;8(3):185-211. doi: 10.1177/108925320400800303. PMID 15375480
- [Result] Zarbock A, Mueller E, Netzer S, Gabriel A, Feindt P, Kindgen-Milles D. Prophylactic nasal continuous positive airway pressure following cardiac surgery protects from postoperative pulmonary complications: a prospective, randomized, controlled trial in 500 patients. Chest. 2009 May;135(5):1252-1259. doi: 10.1378/chest.08-1602. Epub 2008 Nov 18. PMID 19017864
- [Result] Auriant I, Jallot A, Herve P, Cerrina J, Le Roy Ladurie F, Fournier JL, Lescot B, Parquin F. Noninvasive ventilation reduces mortality in acute respiratory failure following lung resection. Am J Respir Crit Care Med. 2001 Oct 1;164(7):1231-5. doi: 10.1164/ajrccm.164.7.2101089. PMID 11673215
- [Result] Zhu GF, Wang DJ, Liu S, Jia M, Jia SJ. Efficacy and safety of noninvasive positive pressure ventilation in the treatment of acute respiratory failure after cardiac surgery. Chin Med J (Engl). 2013 Dec;126(23):4463-9. PMID 24286408
- [Result] Nishimura M. High-Flow Nasal Cannula Oxygen Therapy in Adults: Physiological Benefits, Indication, Clinical Benefits, and Adverse Effects. Respir Care. 2016 Apr;61(4):529-41. doi: 10.4187/respcare.04577. PMID 27016353
- [Result] Corley A, Caruana LR, Barnett AG, Tronstad O, Fraser JF. Oxygen delivery through high-flow nasal cannulae increase end-expiratory lung volume and reduce respiratory rate in post-cardiac surgical patients. Br J Anaesth. 2011 Dec;107(6):998-1004. doi: 10.1093/bja/aer265. Epub 2011 Sep 9. PMID 21908497
- [Result] Parke R, McGuinness S, Dixon R, Jull A. Open-label, phase II study of routine high-flow nasal oxygen therapy in cardiac surgical patients. Br J Anaesth. 2013 Dec;111(6):925-31. doi: 10.1093/bja/aet262. Epub 2013 Aug 6. PMID 23921199
- [Result] Parke RL, McGuinness SP, Eccleston ML. A preliminary randomized controlled trial to assess effectiveness of nasal high-flow oxygen in intensive care patients. Respir Care. 2011 Mar;56(3):265-70. doi: 10.4187/respcare.00801. Epub 2011 Jan 21. PMID 21255498
- [Result] Stephan F, Barrucand B, Petit P, Rezaiguia-Delclaux S, Medard A, Delannoy B, Cosserant B, Flicoteaux G, Imbert A, Pilorge C, Berard L; BiPOP Study Group. High-Flow Nasal Oxygen vs Noninvasive Positive Airway Pressure in Hypoxemic Patients After Cardiothoracic Surgery: A Randomized Clinical Trial. JAMA. 2015 Jun 16;313(23):2331-9. doi: 10.1001/jama.2015.5213. PMID 25980660
- [Result] Zochios V, Klein AA, Jones N, Kriz T. Effect of High-Flow Nasal Oxygen on Pulmonary Complications and Outcomes After Adult Cardiothoracic Surgery: A Qualitative Review. J Cardiothorac Vasc Anesth. 2016 Oct;30(5):1379-85. doi: 10.1053/j.jvca.2015.12.023. Epub 2015 Dec 18. No abstract available. PMID 26976034
- [Result] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Result] Maggiore SM, Idone FA, Vaschetto R, Festa R, Cataldo A, Antonicelli F, Montini L, De Gaetano A, Navalesi P, Antonelli M. Nasal high-flow versus Venturi mask oxygen therapy after extubation. Effects on oxygenation, comfort, and clinical outcome. Am J Respir Crit Care Med. 2014 Aug 1;190(3):282-8. doi: 10.1164/rccm.201402-0364OC. PMID 25003980
- [Result] Esteban A, Alia I, Gordo F, Fernandez R, Solsona JF, Vallverdu I, Macias S, Allegue JM, Blanco J, Carriedo D, Leon M, de la Cal MA, Taboada F, Gonzalez de Velasco J, Palazon E, Carrizosa F, Tomas R, Suarez J, Goldwasser RS. Extubation outcome after spontaneous breathing trials with T-tube or pressure support ventilation. The Spanish Lung Failure Collaborative Group. Am J Respir Crit Care Med. 1997 Aug;156(2 Pt 1):459-65. doi: 10.1164/ajrccm.156.2.9610109. PMID 9279224
- [Result] Godard S, Herry C, Westergaard P, Scales N, Brown SM, Burns K, Mehta S, Jacono FJ, Kubelik D, Maziak DE, Marshall J, Martin C, Seely AJ. Practice Variation in Spontaneous Breathing Trial Performance and Reporting. Can Respir J. 2016;2016:9848942. doi: 10.1155/2016/9848942. Epub 2016 Mar 29. PMID 27445575
- [Result] 34. Vats, N., Singh, J., & Kalra, S. (2012). Extubation outcome after spontaneous breathing trials with T-tube or pressure support ventilation. Indian Journal of Physiotherapy
- [Result] Wilson RC, Jones PW. A comparison of the visual analogue scale and modified Borg scale for the measurement of dyspnoea during exercise. Clin Sci (Lond). 1989 Mar;76(3):277-82. doi: 10.1042/cs0760277. PMID 2924519
- [Result] Gift AG. Validation of a vertical visual analogue scale as a measure of clinical dyspnea. Rehabil Nurs. 1989 Nov-Dec;14(6):323-5. doi: 10.1002/j.2048-7940.1989.tb01129.x. PMID 2813949
- [Result] Carlsson AM. Assessment of chronic pain. I. Aspects of the reliability and validity of the visual analogue scale. Pain. 1983 May;16(1):87-101. doi: 10.1016/0304-3959(83)90088-X. PMID 6602967
- [Result] Adamis D, Dimitriou C, Anifantaki S, Zachariadis A, Astrinaki I, Alegakis A, Mari H, Tsiatsiotis N. Validation of the Greek version of Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Intensive Crit Care Nurs. 2012 Dec;28(6):337-43. doi: 10.1016/j.iccn.2012.02.003. Epub 2012 Mar 8. PMID 22406251
- [Result] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Result] Lopez MG, Pandharipande P, Morse J, Shotwell MS, Milne GL, Pretorius M, Shaw AD, Roberts LJ 2nd, Billings FT 4th. Intraoperative cerebral oxygenation, oxidative injury, and delirium following cardiac surgery. Free Radic Biol Med. 2017 Feb;103:192-198. doi: 10.1016/j.freeradbiomed.2016.12.039. Epub 2016 Dec 27. PMID 28039082
- [Result] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Result] Pun BT, Devlin JW. Delirium monitoring in the ICU: strategies for initiating and sustaining screening efforts. Semin Respir Crit Care Med. 2013 Apr;34(2):179-88. doi: 10.1055/s-0033-1342972. Epub 2013 May 28. PMID 23716309
- [Result] 43. García, G., Agosta, M., Valencia, P., Mercedes, E., & Sarhane, Y. (2017). Avoiding confusion in high fl ow oxygen therapy concepts, 1-2
- [Result] Corley A, Rickard CM, Aitken LM, Johnston A, Barnett A, Fraser JF, Lewis SR, Smith AF. High-flow nasal cannulae for respiratory support in adult intensive care patients. Cochrane Database Syst Rev. 2017 May 30;5(5):CD010172. doi: 10.1002/14651858.CD010172.pub2. PMID 28555461
- [Result] Fernandez R, Subira C, Frutos-Vivar F, Rialp G, Laborda C, Masclans JR, Lesmes A, Panadero L, Hernandez G. High-flow nasal cannula to prevent postextubation respiratory failure in high-risk non-hypercapnic patients: a randomized multicenter trial. Ann Intensive Care. 2017 Dec;7(1):47. doi: 10.1186/s13613-017-0270-9. Epub 2017 May 2. PMID 28466461
- [Result] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03282552/Prot_SAP_ICF_000.pdf